CLINICAL TRIAL: NCT05791292
Title: Investigation of Pressure Pain Threshold and Hand Grip Strength in Individuals With and Without Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 83116987-658
Record Dates: First submitted 2023-03-15; First posted 2023-03-30 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain
Keywords: Pressure pain threshold; Neck; Neck pain; Hand grip strength; Quality of life
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Case control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients group (Other): To evaluate hand grip strength, neck discomfort, arm, shoulder and hand problems, and overall quality of life.
  Interventions: Other: Evaluation
- Healthy group (Other): To evaluate hand grip strength, neck discomfort, arm, shoulder and hand problems, and overall quality of life.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — To evaluate hand grip strength, neck discomfort, arm, shoulder and hand problems, and overall quality of life.

SUMMARY:
This study will be determined whether the pressure pain threshold and hand grip strength are affected in individuals with neck pain compared to individuals without neck pain.

DETAILED DESCRIPTION:
When the literature is examined, there are studies examining different parameters in different occupations, men and women with neck pain, individuals with cervical disc hernia, and individuals with chronic neck pain. Studies have addressed different parameters that may be associated with neck pain from different perspectives. However, no study was found in which the pressure pain threshold and hand grip strengths were determined and the relationship was examined in individuals with and without chronic neck pain. Therefore, with this study, it will be determined whether the pressure pain threshold and hand grip strength are affected in individuals with neck pain compared to individuals without neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain complaint for more than three months,
* Without any diagnosed chronic disease,
* Have no past or present psychological disorders,
* Individuals who can speak, read and write Turkish.

Exclusion Criteria:

* Having any neurological, psychiatric or cognitive disorder,
* Individuals who cannot speak, read or write Turkish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | 1 day
  A hand dynamometer (Baseline® Digital Smedley Dynamometer) will be used to evaluate hand grip strength. Measurements will be made with the feet on the chair in an upright sitting position without elbow support, with the shoulder joint in adduction, the elbow joint in 90 degrees flexion, and the forearm and wrist in the neutral position. Measurements will be made for both the right side and the left side. During the measurements, 3 separate measurements will be made by giving rest intervals and the average of these measurements will be taken and recorded in kilograms (kg).
Neck disorder | 1 day
  Neck disorders will be assessed with the Neck Bournemouth Questionnaire (NBQ). NBQ consists of 7 questions that examine pain intensity, activities of daily living, social activities, anxiety, emotional aspects of depression, kinesiophobia, and ability to control pain. The items in the questionnaire are specific to patients with neck pain, and each question evaluates a different parameter. A high score indicates a high degree of discomfort. The Turkish version of the NBQ has been proven to be valid and reliable.
Arm, shoulder, and hand problems | 1 day
  Arm, shoulder, and hand problems will be assessed with the Disabilities of the Arm, Shoulder, and Hand (DASH). DASH is an abbreviated version of DASH to measure physical function and symptoms in patients with upper extremity musculoskeletal disorders. Answers are given on a scale of one to five, and each question is scored from 1 to 5. Scores on the three subscales of the DASH disability/symptom scale, the work scale, and the sports/performing arts scale all range from 0 (no disability) to 100 (most severe disability). The Turkish version of DASH has been reported to be valid and reliable.
General quality of life | 1 day
  The Nottingham Health Profile (NHP) is a general quality of life questionnaire that measures a person's perceived health problems and the extent to which these problems affect normal daily activities. The NHP consists of 38 items. Questions are answered as 'yes' or 'no'. The questionnaire assesses six parameters related to health status. These parameters are; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items), and emotional reactions (9 items). Each sub-parameter is scored between 0-100. 0 indicates best health, and 100 indicates worst health. The total NHP score is derived from the sum of the subscores.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)